CLINICAL TRIAL: NCT06212921
Title: Biomarkers In Prediction of Acute Mesenteric Ischaemia: a Prospective Multicentre Study (BIPAMI Study)
Brief Title: Biomarkers in Prediction of AMI
Acronym: BIPAMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Annika Reintam Blaser, Associate Professor, University of Tartu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BIPAMI study
Record Dates: First submitted 2024-01-04; First posted 2024-01-19 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Acute Mesenteric Ischemia

STUDY DESIGN:
Intervention Model Description: Sequential blood samples will be collected from study subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with suspicion of acute mesenteric ischaemia (Other): Bolld samples is the only intervention. All patients with suspicion of AMI will be included and blood samples collected
  Interventions: Diagnostic Test: Sequential blood samples

INTERVENTIONS:
Diagnostic Test: Sequential blood samples — Sequential blood samples for diagnostic tests is the only intervention in thei study

SUMMARY:
Current study will be undertaken to identify combinations of biomarkers that can reliably identify acute mesenteric ischaemia (AMI) and distinguish between non-transmural and transmural ischaemia. Different combinations of biomarkers for different sub-types and severity of AMI, and different time points of measurement after onset of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Initial decision in favour of further diagnostics of mesenteric ischaemia

Exclusion Criteria:

* Age <18 years
* Consent declined by patient or next of kin (delayed consent)
* Chronic mesenteric ischaemia without an acute event
* Immediate decision for withdrawal of further diagnostics and active treatment
* Referral from another hospital with already established diagnosis of AMI
* AMI diagnosed at surgery without previously having been considered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of correctly predicted cases of acute mesenteric ischaemia | 10 months
  Rate of correctly predicted cases of Acute mesenteric ischaemia using different biomarkers

CONTACTS AND LOCATIONS:
Locations (2):
- Tartu University Hospital, Tartu, Estonia
- Lucerne Cantonal Hospital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tamme K, Acosta S, Biloslavo A, Bjorck M, Casian D, Damaskos D, Forbes A, Kase K, Kisand K, Lakbar I, Mihnovits V, Murruste M, Mandul M, Nuzzo A, Padar M, Starkopf J, Visconti D, Reintam Blaser A. Biomarkers In Prediction of Acute Mesenteric Ischaemia: a prospective multicentre study (BIPAMI study): a study protocol. BMC Surg. 2024 Jul 3;24(1):201. doi: 10.1186/s12893-024-02491-3. PMID 38961419